CLINICAL TRIAL: NCT02909517
Title: The Role of Inflammation in Ocular Tumours
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 14-416
Record Dates: First submitted 2016-09-16; First posted 2016-09-21 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Ocular Melanoma
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (5):
- Choroidal nevus: Requires distinction from melanoma through diagnostic testing (low-risk features)
  Interventions: Other: cSLO imaging
- Choroidal indeterminate melanocytic lesion: Requires diagnostic testing for identification and distinction from nevus and melanoma (high-risk features)
  Interventions: Other: cSLO imaging
- Choroidal melanoma: Requires confirmation of diagnosis and evaluation for potential metatstases
  Interventions: Other: cSLO imaging
- Suspected metastatic tumour: Requires identification of primary tumour (ie, primary tumour elsewhere)
  Interventions: Other: cSLO imaging
- Locally treated ocular tumour: Requires followup to evaluate response to treatment and potential change or repeat therapy
  Interventions: Other: cSLO imaging

INTERVENTIONS:
Other: cSLO imaging

SUMMARY:
This prospective, non-therapeutic study will determine whether a novel imaging technique can identify presumptive tumour associated macrophages (TAMs) in patients with ocular tumours.

The investigators will evaluate 5 groups:

1. Choroidal nevus
2. Choroidal indeterminate melanocytic lesion
3. Choroidal melanoma
4. Suspected metastatic tumour (ie, primary tumour elsewhere)
5. Locally treated ocular tumours

ELIGIBILITY:
Inclusion Criteria:

Any tentative clinical diagnosis of:

1. Choroidal nevus (low-risk features):
2. Choroidal indeterminate melanocytic lesion (high-risk features)
3. Choroidal melanoma
4. Suspected metastatic tumour (ie, primary tumour elsewhere)
5. Locally treated ocular tumours

Note that a patient can enroll in this study twice, once before treatment and once after, provided that at least one month has passed since initiation of treatment. This patient will count twice (ie, once in each of two study arms)

Male and female age 18 years and older Ability to provide informed consent

Exclusion Criteria:

* Allergy to angiography dye
* Cases that do not meet the above criteria for tumor size will be ineligible to participate in the study.
* Patients not able to provide consent for the study.
* Patients with a poor view of the fundus due to cataract or vitreous hemorrhage.
* Patients < 18 years of age. Any concurrent unrelated eye diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential study subjects will be identified from within the circle of care of the attending physicians. Subjects must be 18 years of age or older, be able to understand the study protocol, and provide informed consent. They must be able to attend all three visits
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Identification of macrophages | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Shelley Boyd, MD, Principal Investigator — Unity Health Toronto
Locations (2):
- Canada (2):
  - St Michael's Hospital, Toronto, Ontario
  - Princess Margaret Cancer Centre, Ontario, Toronto, Ontario